CLINICAL TRIAL: NCT02691819
Title: Short Term and Long Term Effects of Single Stent and Embedded Balloon Angioplasty in the Treatment of Coronary Bifurcation Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ZhangWenduo (Other Government)
Responsible Party: Sponsor-Investigator, ZhangWenduo, Beijing Hospital, Beijing Hospital
Organization: Beijing Hospital (Other Government)
Other Study IDs: BeijingHZWD001
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-01

CONDITIONS: Percutaneous Coronary Intervention
Keywords: jailed-balloon technique
MeSH Terms: interventions — Stents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months

INTERVENTIONS:
Device: single stent and embedded balloon angioplasty

SUMMARY:
At the same time in the side branch stent expansion vessels were embedded and balloon dilatation technique in for Medina1.1.1 type, 1.0.1 type or 0.1.1 type lesions of interventional therapy for bifurcation lesions, the PCI preoperative and postoperative 6 h, 24h of all patients were at least three times ECG and assay of creatine kinase isoenzyme (CK-MB) and cardiac troponin T (TNT data analysis); immediately after operation and nine months after surgery, coronary angiography, quantitative coronary angiography, evaluation of each main branch and side branch of the lesion degree of stenosis (determination of bifurcation angle, reference vessel diameter, vessel diameter, minimum) and TIMI flow grade; using 256 slice spiral CT scanner to scan each main branch lesion and evaluation a side branch stenosis (determination of bifurcation angle, reference vessel diameter, vessel diameter, minimum). All patients were followed up for 1 months, 6 months, and 9 months follow-up. Cardiovascular events included total cause of death, cardiac death, total re hospitalization rate, recurrent myocardial infarction or unstable angina.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria: selected patients aged 18-80 years of intervention in patients. Baseline characteristics of the patients with screening and recorded by a case by coronary artery angiography of each coronary bifurcation lesions according to the Medina classification method to classify, only select the 1.1.1 type, type 1.0.1 or 0.1.1 type III lesions, a total of 80, respectively, of the type of bifurcation lesions, the random number method lesions were divided into according to the ratio of 1:3 established traditional surgical PCI group 20 lesions and a new operative method for 60 lesions group and interventional therapy. All patients who were involved in the treatment before treatment (sign) or their family members agreed to and signed informed consent. All patients were pre evaluated for long-term oral aspirin (100 mg/, once daily) and clopidogrel (75 mg/ times a day) for at least 1 years

Exclusion Criteria:

Be of aspirin or clopidogrel allergy or intolerance are; the illness history of stroke or visceral hemorrhage within six months; serious liver disease and (or) coagulation abnormality; with antiplatelet treatment contraindications or recently proposed surgical person; valvular heart disease, cardiomyopathy, myocarditis, congenital heart disease, peripheral vascular disease, infection endocarditis; late kidney function not whole, tumor and chronic heart failure seriously affect the short-term prognosis of disease.Patients unable to complete follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Baseline characteristics of the patients with screening and recorded by a case by coronary artery angiography of each coronary bifurcation lesions according to the Medina classification method to classify, only select the 1.1.1 type, type 1.0.1 or 0.1.1 type III lesions,.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
MACE | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhang Wenduo, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Sharma SK, Sweeny J, Kini AS. Coronary bifurcation lesions: a current update. Cardiol Clin. 2010 Feb;28(1):55-70. doi: 10.1016/j.ccl.2009.10.001. PMID 19962049
- [Background] Murasato Y, Hikichi Y, Nakamura S, Kajiya F, Iwasaki K, Kinoshita Y, Yamawaki M, Shinke T, Yamada S, Yamashita T, Choo GH, Nam CW, Kim YH, Jepson N, Ferenc M. Recent perspective on coronary bifurcation intervention: statement of the "Bifurcation Club in KOKURA". J Interv Cardiol. 2010 Aug;23(4):295-304. doi: 10.1111/j.1540-8183.2010.00570.x. PMID 20718905
- [Background] Stankovic G, Lefevre T, Chieffo A, Hildick-Smith D, Lassen JF, Pan M, Darremont O, Albiero R, Ferenc M, Finet G, Adriaenssens T, Koo BK, Burzotta F, Louvard Y; European Bifurcation Club. Consensus from the 7th European Bifurcation Club meeting. EuroIntervention. 2013 May 20;9(1):36-45. doi: 10.4244/EIJV9I1A7. No abstract available. PMID 23552575
- [Background] von Korn H, Stefan V, van Ewijk R, Chakraborty K, Sanwald B, Andel R, Hemker J, Hink U, Ohlow M, Lauer B, Muenzel T. Treatment of coronary bifurcation lesions: stent-covering of the side branch with and without PCI of the side branch: a retrospective analysis of all consecutive patients. BMC Cardiovasc Disord. 2013 Apr 4;13:27. doi: 10.1186/1471-2261-13-27. PMID 23557395
- [Background] Poorhosseini HR, Kassaian SE, Hosseini SK, Fotoohi M, Salarifar M, Alidoosti M, Sharafi A, Nozari Y, Nematipour E, Aghajani H, Haji Zeinali AM, Amirzadegan A, Babapour B, Seyed Mohammad Zadeh MH. Impact of side-branch flow in coronary bifurcation intervention. J Tehran Heart Cent. 2012 Aug;7(3):100-5. Epub 2012 Aug 31. PMID 23304177
- [Background] Maeng M, Holm NR, Erglis A, Kumsars I, Niemela M, Kervinen K, Jensen JS, Galloe A, Steigen TK, Wiseth R, Narbute I, Gunnes P, Mannsverk J, Meyerdierks O, Rotevatn S, Nikus K, Vikman S, Ravkilde J, James S, Aaroe J, Ylitalo A, Helqvist S, Sjogren I, Thayssen P, Virtanen K, Puhakka M, Airaksinen J, Christiansen EH, Lassen JF, Thuesen L; Nordic-Baltic Percutaneous Coronary Intervention Study Group. Long-term results after simple versus complex stenting of coronary artery bifurcation lesions: Nordic Bifurcation Study 5-year follow-up results. J Am Coll Cardiol. 2013 Jul 2;62(1):30-4. doi: 10.1016/j.jacc.2013.04.015. Epub 2013 May 1. PMID 23644088
- [Background] Kang SJ, Kim WJ, Lee JY, Park DW, Lee SW, Kim YH, Lee CW, Mintz GS, Park SW, Park SJ. Hemodynamic impact of changes in bifurcation geometry after single-stent cross-over technique assessed by intravascular ultrasound and fractional flow reserve. Catheter Cardiovasc Interv. 2013 Dec 1;82(7):1075-82. doi: 10.1002/ccd.24956. Epub 2013 Aug 1. PMID 23592548
- [Background] Steigen TK, Maeng M, Wiseth R, Erglis A, Kumsars I, Narbute I, Gunnes P, Mannsverk J, Meyerdierks O, Rotevatn S, Niemela M, Kervinen K, Jensen JS, Galloe A, Nikus K, Vikman S, Ravkilde J, James S, Aaroe J, Ylitalo A, Helqvist S, Sjogren I, Thayssen P, Virtanen K, Puhakka M, Airaksinen J, Lassen JF, Thuesen L; Nordic PCI Study Group. Randomized study on simple versus complex stenting of coronary artery bifurcation lesions: the Nordic bifurcation study. Circulation. 2006 Oct 31;114(18):1955-61. doi: 10.1161/CIRCULATIONAHA.106.664920. Epub 2006 Oct 23. PMID 17060387
- [Background] Hildick-Smith D, Lassen JF, Albiero R, Lefevre T, Darremont O, Pan M, Ferenc M, Stankovic G, Louvard Y; European Bifurcation Club. Consensus from the 5th European Bifurcation Club meeting. EuroIntervention. 2010 May;6(1):34-8. No abstract available. PMID 20542795